CLINICAL TRIAL: NCT03708211
Title: A Phase 1, Open-Label Study to Assess the Relative Bioavailability, Effect of Food, and Gastric pH Modification on the Pharmacokinetics of TAK-931 in Patients With Advanced Solid Tumors
Brief Title: A Study to Assess the Relative Bioavailability, Effect of Food, and Gastric Potential Hydrogen (pH) Modification on the Pharmacokinetics (PK) of TAK-931 in Participants With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: TAK-931-1003; 2017-004629-34 (EudraCT Number); U1111-1214-4266 (Registry Identifier: WHO); NL66709.091.18 (Registry Identifier: Netherlands (CCMO))
Record Dates: First submitted 2018-10-12; First posted 2018-10-17 (Actual); Results first posted 2020-12-29 (Actual); Last update posted 2020-12-29 (Actual); Status verified 2020-12

CONDITIONS: Neoplasms, Advanced Solid
Keywords: Drug Therapy
MeSH Terms: conditions — Neoplasms | interventions — simurosertib; Esomeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Part1: TAK-931 80 mg PIC + TAK-931 80 mg Tablet (Experimental): TAK-931 80 milligram (mg), PIC, orally, once on Day 1 Cycle 0 (16-day treatment cycle), followed by TAK-931 80 mg, tablet, orally, once on Day 3 Cycle 0, further followed by TAK-931 50 mg, PIC, orally, once daily from Day 5 to Day 16 Cycle 0. Participants will receive TAK-931 50 mg PIC, orally, once daily for up to 14 days in 21-day treatment cycles until progressive disease (PD), or unacceptable toxicity or any treatment discontinuation is determined.
  Interventions: Drug: TAK-931 PIC; Drug: TAK-931 Tablet
- Part1: TAK-931 80 mg Tablet + TAK-931 80 mg PIC (Experimental): TAK-931 80 mg, tablet, orally, once on Day 1 of Cycle 0 (16-day treatment cycle), followed by TAK-931 80 mg, PIC, orally, once on Day 3 Cycle 0, further followed by TAK-931 50 mg, PIC, orally, once daily from Day 5 to Day 16 Cycle 0. Participants will receive TAK-931 50 mg PIC, orally, once daily for up to 14 days in 21-day treatment cycles until PD, or unacceptable toxicity or any treatment discontinuation is determined.
  Interventions: Drug: TAK-931 PIC; Drug: TAK-931 Tablet
- Part 2: TAK-931 Fed + TAK-931 Fasted + Esomeprazole 40 mg (Experimental): TAK-931 tablet, orally, once under fed state on Day 1 Cycle 0 (22-day treatment cycle), followed by TAK-931 tablet, orally, once under fasted state on Day 3 Cycle 0, further followed by esomeprazole 40 mg, tablet, orally, once daily from Day 5 to Day 13 Cycle 0 and TAK-931 tablet, orally, once on Day 12, Day 14 to Day 22. Participants will receive TAK-931 tablets, orally, once daily for up to 14 days in 21-day treatment cycles until PD, unacceptable toxicity or any treatment discontinuation is determined. Dose of TAK-931 in Part 2 will be determined based on relative bioavailability data available from Part 1 of the study.
  Interventions: Drug: TAK-931 Tablet; Drug: Esomeprazole
- Part 2: TAK-931 Fasted + TAK-931 Fed + Esomeprazole 40 mg (Experimental): TAK-931 tablet, orally, once under fasted state on Day 1 Cycle 0 (22-day treatment cycle), followed by TAK-931 tablet, orally, once under fed state on Day 3 Cycle 0, further followed by esomeprazole 40 mg, tablet, orally, once daily from Day 5 to Day 13 Cycle 0 and TAK-931 tablet, orally, once on Day 12, Day 14 to Day 22. Participants will receive TAK-931 tablets, orally, once daily for up to 14 days in 21-day treatment cycles until PD, unacceptable toxicity or any treatment discontinuation is determined. Dose of TAK-931 in Part 2 will be determined based on relative bioavailability data available from Part 1 of the study.
  Interventions: Drug: TAK-931 Tablet; Drug: Esomeprazole

INTERVENTIONS:
Drug: TAK-931 PIC — TAK-931 PICs.
  Arms: Part1: TAK-931 80 mg PIC + TAK-931 80 mg Tablet; Part1: TAK-931 80 mg Tablet + TAK-931 80 mg PIC
Drug: TAK-931 Tablet — TAK-931 Tablets.
Drug: Esomeprazole — Esomeprazole Tablets.
  Arms: Part 2: TAK-931 Fasted + TAK-931 Fed + Esomeprazole 40 mg; Part 2: TAK-931 Fed + TAK-931 Fasted + Esomeprazole 40 mg

SUMMARY:
The purpose of this study is to estimate the relative bioavailability of TAK-931 tablets in reference to powder-in capsule (PIC) and to assess the effect of food and esomeprazole on the pharmacokinetics (PK) of TAK-931 as a tablet.

DETAILED DESCRIPTION:
The drug being tested in this study is called TAK-931. TAK 931 is being tested to treat participants who have advanced solid tumors. This study will look at relative bioavailability, effect of food and gastric pH modification on the PK of TAK-931.

The study will enroll approximately 44 participants. The study will be conducted in 2 parts: Part 1 and Part 2. In Part 1 and Part 2, participants will be randomly assigned (by chance, like flipping a coin) in a crossover design. In Part 1, participants will be assigned to 1 of the 2 following treatment sequences:

* TAK-931 80 mg PIC + TAK-931 80 mg Tablet
* TAK-931 80 mg Tablet + TAK-931 80 mg PIC

Part 2 of the study will be initiated, once the preliminary PK data from Part 1 is available to determine the relative bioavailability of the tablet formulation in reference to PIC and to calculate the single dose of TAK-931 tablet to be used in Part 2.In Part 2, participants will be assigned to 1 of the 2 following treatment sequences:

* TAK-931 TBD Fed + TAK-931 TBD Fasted
* TAK-931 TBD Fasted + TAK-931 TBD Fed

This multi-center trial will be conducted in the Netherlands. The overall time to participate in this study is approximately 2 years. Participants will make multiple visits to the clinic and will be contacted for approximately 30 days after receiving their last dose of study drug or until the start of subsequent anticancer therapy, whichever occurs first for a follow up assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Adult participants with histologically or cytologically confirmed metastatic or locally advanced or metastatic solid tumors for whom there is no available standard treatment with proven survival benefit, this therapy is not indicated, or it is refused by the participant. Based on the nonclinical data, the following indications may have a higher probability of clinical benefit: high-grade serous ovarian cancer, uterine carcinosarcoma, squamous esophageal cancer, squamous non-small cell lung carcinoma (NSCLC), rectal adenocarcinoma, and in general tumors with known tumor protein 53 (TP53) gene mutations. For any of these preferred indications, participants should have exhausted standard therapeutic options with a proven survival benefit.
2. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1.
3. Recovered to Grade 1 or baseline from all toxic effects of previous therapy (except alopecia or neuropathy).
4. Suitable venous access for the study-required blood sampling including PK and pharmacodynamic sampling.
5. Must have a radiographically or clinically evaluable tumor, but measurable disease as defined by RECIST v1.1 is not required for participation in this study.

Exclusion Criteria:

1. Participants who require continuous use of proton pump inhibitors (PPIs) or histamine-2 (H2) receptor antagonists and participants who are taking PPIs within 5 days before the first dose of study drug.
2. Treatment with clinically significant enzyme inducers, such as phenytoin, carbamazepine, enzalutamide, mitotane, ritonavir, rifampin, or St John's wort within 14 days before the first dose of study drug.
3. With treated brain metastases are eligible if there is no evidence of progression for at least 4 weeks after central nervous system-directed treatment, as ascertained by clinical examination and brain imaging (magnetic resonance imaging [MRI] or CT) during the screening period.
4. Part 2 only: known hypersensitivity to PPIs (example, angioedema or anaphylaxis have occurred).
5. Part 2 only: not being able or willing to take one high fat breakfast as indicated in the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-03-28 (Actual); Primary Completion 2019-12-03 (Actual); Study Completion 2019-12-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Millennium Pharmaceuticals, Inc.
Locations (4):
- Netherlands (4):
  - Radboud University Medical Center, Department of Medical Oncology, Nijmegen, Gelderland
  - Netherlands Cancer Institute - Antoni van Leeuwenhoek, Department of Medical Oncology, Amsterdam, North Holland
  - Leiden University Medical Center, Department of Clinical Oncology, Leiden, South Holland
  - Erasmus MC Cancer Institute, Department of Internal Oncology, Rotterdam, South Holland

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- [Derived] Steeghs N, Pruis M, van Herpen C, Lu V, Redman J, Zhou X. A phase 1 open-label study to assess the relative bioavailability of TAK-931 tablets in reference to powder-in-capsule in patients with advanced solid tumors. Invest New Drugs. 2023 Feb;41(1):53-59. doi: 10.1007/s10637-022-01318-3. Epub 2022 Nov 21. PMID 36409435

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at investigative sites in the Netherlands from 28 March 2019 to 03 December 2019.
Pre-assignment Details: Participants with advanced solid tumors were enrolled in 2-part cross-over design study to receive 1 of 2 treatment sequences in Part 1: TAK-931 80 mg PIC + TAK-931 80 mg tablet (Sequence A) or TAK-931 80 mg tablet + TAK-931 80 mg PIC (Sequence B). Part 2 of the study was not conducted due to the business decision, which was unrelated to safety.
Groups:
- Part 1, Sequence A: TAK-931 80 mg PIC + TAK-931 80 mg Tablet: TAK-931 80 milligram (mg), powder in capsule (PIC), orally, once on Day 1, followed by TAK-931 80 mg tablet, orally, once on Day 3, further followed by TAK-931 50 mg PIC, orally, once daily from Days 5 to 16 in Cycle 0 (16-day treatment cycle), followed by a 7-day rest period, further followed by TAK-931 50 mg PIC, orally, once daily for up to 14 days in Cycle 1, followed by a 7-day rest period in 21-day treatment cycles, until progressive disease (PD), or unacceptable toxicity or any treatment discontinuation is determined.
- Part 1, Sequence B: TAK-931 80 mg Tablet + TAK-931 80 mg PIC: TAK-931 80 mg, tablet, orally, once on Day 1, followed by TAK-931 80 mg PIC, orally, once on Day 3, further followed by TAK-931 50 mg PIC, orally, once daily from Day 5 to Day 16 in Cycle 0 (16-day treatment cycle), followed by a 7-day rest period, further followed by TAK-931 50 mg PIC, orally, once daily for up to 14 days in Cycle 1, followed by a 7-day rest period in 21-day treatment cycles until PD, or unacceptable toxicity or any treatment discontinuation is determined.
Period: Overall Study
Arm/Group | Part 1, Sequence A: TAK-931 80 mg PIC + TAK-931 80 mg Tablet | Part 1, Sequence B: TAK-931 80 mg Tablet + TAK-931 80 mg PIC
Started | 12 | 8
Completed | 0 | 0
Not Completed | 12 | 8
Not completed — Progressive Disease | 10 | 7
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Other | 2 | 0

BASELINE CHARACTERISTICS:
Population: The safety set included all participants who received any amount of study drug.
Groups:
- Part 1, Sequence A: TAK-931 80 mg PIC + TAK-931 80 mg Tablet: TAK-931 80 mg, PIC, orally, once on Day 1, followed by TAK-931 80 mg tablet, orally, once on Day 3, further followed by TAK-931 50 mg PIC, orally, once daily from Days 5 to 16 in Cycle 0 (16-day treatment cycle), followed by a 7-day rest period, further followed by TAK-931 50 mg PIC, orally, once daily for up to 14 days in Cycle 1, followed by a 7-day rest period in 21-day treatment cycles, until PD, or unacceptable toxicity or any treatment discontinuation is determined.
- Total: Total of all reporting groups
Arm/Group | Part 1, Sequence A: TAK-931 80 mg PIC + TAK-931 80 mg Tablet | Part 1, Sequence B: TAK-931 80 mg Tablet + TAK-931 80 mg PIC | Total
Number analyzed (Participants) | 12 | 8 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.6 (9.36) | 57.6 (12.69) | 60.6 (10.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 8
  Male | 8 | 4 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 1 | 0 | 1
  Unknown or Not Reported | 11 | 8 | 19
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 3 | 2 | 5
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 9 | 6 | 15
Region of Enrollment [Count of Participants; unit: Participants]
  Netherlands | 12 | 8 | 20
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilogram per square meter (kg/m^2)] | 26.56 (2.165) | 26.50 (5.292) | 26.53 (3.610)

OUTCOME MEASURES:

1. Primary Outcome: Part 1, Cmax: Maximum Observed Plasma Concentration for TAK-931 Tablets in Reference to PIC
Time Frame: Cycle 0 Days 1 and 3 pre-dose and at multiple time points (up to 48 hours) post-dose (Cycle 0 length is equal to [=] 16 days)
Population: The pharmacokinetic (PK) set included all participants who completed the protocol-specified dosing and had sufficient plasma TAK-931 concentration-time data to reliably estimate the PK parameter.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Groups:
- TAK-931 80 mg PIC: TAK-931 80 mg, PIC, orally, once, on Day 1 or Day 3 of Cycle 0, further followed by TAK-931 50 mg PIC, orally, once daily from Day 5 to Day 16 in Cycle 0 (16-day treatment cycle), followed by a 7-day rest period, further followed by TAK-931 50 mg PIC, orally, once daily for up to 14 days in Cycle 1, followed by a 7-day rest period in 21-day treatment cycles until PD, or unacceptable toxicity or any treatment discontinuation is determined.
- TAK-931 80 mg Tablet: TAK-931 80 mg, tablet, orally, once, on Day 1 or Day 3 of Cycle 0, further followed by TAK-931 50 mg PIC, orally, once daily from Day 5 to Day 16 in Cycle 0 (16-day treatment cycle), followed by a 7-day rest period, further followed by TAK-931 50 mg PIC, orally, once daily for up to 14 days in Cycle 1, followed by a 7-day rest period in 21-day treatment cycles until PD, or unacceptable toxicity or any treatment discontinuation is determined.
Arm/Group | TAK-931 80 mg PIC | TAK-931 80 mg Tablet
Number analyzed (Participants) | 20 | 20
nanogram per milliliter (ng/mL) | 251.45 (41.91) | 270.09 (36.44)
Statistical Analysis 1: Comparison: TAK-931 80 mg PIC vs TAK-931 80 mg Tablet; Following log-transformation, PK parameters were analyzed by analysis of variance (ANOVA) fitting terms for treatment group, sequence and period. Participants within sequence were treated as a random effect. The obtained point estimates and adjusted 90 percent (%) confidence intervals (CIs) for difference in treatment were exponentially back transformed to provide point and confidence interval estimates for the ratios of interest appropriately; Test type: Other; Ratio of geometric mean = 0.9359, 90% CI 2-sided [0.8084 to 1.0835]

2. Primary Outcome: Part 1, AUClast: Area Under the Plasma Concentration-time Curve From Time 0 to the Time of the Last Quantifiable Concentration for TAK-931 Tablets in Reference to PIC
Time Frame: Cycle 0 Days 1 and 3 pre-dose and at multiple time points (up to 48 hours) post-dose (Cycle 0 length = 16 days)
Population: The PK set included all participants who completed the protocol-specified dosing and had sufficient plasma TAK-931 concentration-time data to reliably estimate the PK parameter.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*nanogram per milliliter (h*ng/mL)
Arm/Group | TAK-931 80 mg PIC | TAK-931 80 mg Tablet
Number analyzed (Participants) | 20 | 20
hour*nanogram per milliliter (h*ng/mL) | 1869.0329 (44.7484) | 1898.9016 (45.2980)
Statistical Analysis 1: Comparison: TAK-931 80 mg PIC vs TAK-931 80 mg Tablet; Following log-transformation, PK parameters were analyzed by ANOVA fitting terms for treatment group, sequence and period. Participants within sequence were treated as a random effect. The obtained point estimates and adjusted 90% CIs for difference in treatment were exponentially back transformed to provide point and confidence interval estimates for the ratios of interest appropriately; Test type: Other; Ratio of geometric mean = 1.0036, 90% CI 2-sided [0.8992 to 1.1201]

3. Primary Outcome: Part 1, AUC∞: Area Under the Plasma Concentration-time Curve From Time 0 to Infinity for TAK-931 Tablets in Reference to PIC
Time Frame: Cycle 0 Days 1 and 3 pre-dose and at multiple time points (up to 48 hours) post-dose (Cycle 0 length = 16 days)
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | TAK-931 80 mg PIC | TAK-931 80 mg Tablet
Number analyzed (Participants) | 20 | 20
h*ng/mL | 1901.1447 (44.6999) | 1925.8648 (45.2966)
Statistical Analysis 1: Comparison: TAK-931 80 mg PIC vs TAK-931 80 mg Tablet; [analysis description as in outcome 2, analysis 1]; Test type: Other; Ratio of geometric mean = 1.0071, 90% CI 2-sided [0.9033 to 1.1227]

4. Secondary Outcome: Part 1, Tmax: Time to Reach the Maximum Plasma Concentration (Cmax) for TAK-931 as PIC and Tablets
Time Frame: Cycle 0 Days 1 and 3 pre-dose and at multiple time points (up to 48 hours) post-dose (Cycle 0 length = 16 days)
Population: as for outcome 2
Measure: Median (Full Range); unit: hour
Arm/Group | TAK-931 80 mg PIC | TAK-931 80 mg Tablet
Number analyzed (Participants) | 20 | 20
hour | 1.6830 [0.917 to 4.117] | 1.9830 [0.483 to 4.033]

5. Secondary Outcome: Part 1, CL/F: Oral Clearance for TAK-931
Time Frame: Cycle 0 Days 1 and 3 pre-dose and at multiple time points (up to 48 hours) post-dose (Cycle 0 length = 16 days)
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liter per hour (L/h)
Arm/Group | TAK-931 80 mg PIC | TAK-931 80 mg Tablet
Number analyzed (Participants) | 20 | 20
liter per hour (L/h) | 42.0799 (44.6999) | 41.5397 (45.2966)

6. Secondary Outcome: Part 1, T1/2z: Terminal Disposition Phase Half-life for TAK-931
Time Frame: Cycle 0 Days 1 and 3 pre-dose and at multiple time points (up to 48 hours) post-dose (Cycle 0 length = 16 days)
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour
Arm/Group | TAK-931 80 mg PIC | TAK-931 80 mg Tablet
Number analyzed (Participants) | 20 | 20
hour | 7.3250 (25.4121) | 7.3683 (18.6369)

7. Secondary Outcome: Part 1: Overall Response Rate (ORR)
Description: ORR was defined as the percentage of participants achieving complete response (CR) and partial response (PR) as assessed by Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1), CR was defined as disappearance of all lesions, PR was defined as at least a 30% decrease in the sum of the longest diameter (LD) of lesions, taking as reference the baseline sum LD.
Time Frame: Baseline up to 8 months
Population: The response-evaluable population included participants who received at least 1 dose of study drug, had measurable disease at baseline, and had at least 1 postbaseline response. As planned, efficacy data was collected and analyzed as per sequence and in accordance with the study design.
Measure: Number; unit: percentage of participants
Arm/Group | Part 1, Sequence A: TAK-931 80 mg PIC + TAK-931 80 mg Tablet | Part 1, Sequence B: TAK-931 80 mg Tablet + TAK-931 80 mg PIC
Number analyzed (Participants) | 11 | 8
percentage of participants | 0 | 0

8. Secondary Outcome: Part 1: Progression-free Survival (PFS)
Description: PFS was defined as the time from the date of randomization to the date of first documentation of PD or death due to any cause, whichever occured first. Per RECIST V1.1, PD was defined as at least a 20% increase in the SoD (Sum of Diameters) of target lesions, taking as a reference the smallest (nadir) SoD since (and including) baseline. In addition to the relative increase of 20%, the SoD must also demonstrate an absolute increase of at least 5 millimeter (mm).
Time Frame: From the date of randomization to the date of first documentation of PD or death due to any cause, whichever occurred first (up to 8 months)
Population: The safety set included all participants who received any amount of study drug. As planned, efficacy data was collected and analyzed as per sequence and in accordance with the study design.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Part 1, Sequence A: TAK-931 80 mg PIC + TAK-931 80 mg Tablet | Part 1, Sequence B: TAK-931 80 mg Tablet + TAK-931 80 mg PIC
Number analyzed (Participants) | 12 | 8
months | 1.9 [1.7 to 2.8] | 2.0 [1.4 to 3.6]

9. Secondary Outcome: Part 1: Disease Control Rate (DCR)
Description: DCR was defined as the percentage of participants with CR, PR plus stable disease (SD) greater than or equal to (>=) 1 post baseline computed tomography (CT) scan evaluation from treatment initiation to qualify for DCR. Per RECIST v 1.1, CR was defined as disappearance of all lesions. PR was defined as at least a 30% decrease in the sum of the LD of lesions, taking as reference the baseline sum LD. PD was defined as at least a 20% increase in the SoD of target lesions, taking as a reference the smallest (nadir) SoD since (and including) baseline. In addition to the relative increase of 20%, the SoD must also demonstrate an absolute increase of at least 5 mm. SD was defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum LD since the treatment started.
Time Frame: Baseline up to 8 months
Population: as for outcome 7
Measure: Number; unit: percentage of participants
Arm/Group | Part 1, Sequence A: TAK-931 80 mg PIC + TAK-931 80 mg Tablet | Part 1, Sequence B: TAK-931 80 mg Tablet + TAK-931 80 mg PIC
Number analyzed (Participants) | 11 | 8
percentage of participants | 18.2 | 25.0

10. Secondary Outcome: Part 1: Duration of Response (DOR)
Description: DOR was defined as the time from the date of first documentation of a response to the date of first documentation of PD. Per RECIST v1.1, CR was defined as disappearance of all lesions, PR was defined as at least a 30% decrease in the sum of the LD of lesions, taking as reference the baseline sum LD. PD was defined as at least a 20% increase in the SoD of target lesions, taking as a reference the smallest (nadir) SoD since (and including) baseline. In addition to the relative increase of 20%, the SoD must also demonstrate an absolute increase of at least 5 mm.
Time Frame: From the date of first documentation of a response to the date of first documentation of PD ( up to 8 months)
Population: The response-evaluable population included participants who received at least 1 dose of study drug, had measurable disease at baseline, and had at least 1 postbaseline response. Here overall number of participants "N" are those who had CR or PR. As planned, efficacy data was collected and analyzed as per sequence and in accordance with the study design.
Arm/Group | Part 1, Sequence A: TAK-931 80 mg PIC + TAK-931 80 mg Tablet | Part 1, Sequence B: TAK-931 80 mg Tablet + TAK-931 80 mg PIC
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Part 1: Percentage of Participants With Serious Adverse Events (SAEs), Treatment-emergent Adverse Events (TEAEs), and TEAEs Leading to Discontinuation or Dose Modification
Time Frame: From the start of the study drug up to Day 30 after the last dose of study drug (up to 8 months)
Population: The safety set included all participants who received any amount of study drug. As planned, safety data was collected and analyzed as per sequence and in accordance with the study design.
Measure: Number; unit: percentage of participants
Arm/Group | Part 1, Sequence A: TAK-931 80 mg PIC + TAK-931 80 mg Tablet | Part 1, Sequence B: TAK-931 80 mg Tablet + TAK-931 80 mg PIC
Number analyzed (Participants) | 12 | 8
percentage of participants
  SAEs | 16.7 | 25.0
  TEAEs | 91.7 | 100
  TEAEs Leading to Discontinuation or Dose Modification | 8.3 | 0

12. Secondary Outcome: Part 1: Percentage of Participants With Grade 3 or Higher TEAEs
Description: An AE was defined as any untoward medical occurrence in a participant who has enrolled in a study; it does not necessarily have a causal relationship with this treatment. A treatment-emergent adverse event (TEAE) was defined as an adverse event with an onset that occurs after receiving study drug. A severity grade was defined by the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) Version 5.0. As per NCI-CTCAE, Grade 1 scales as Mild; Grade 2 scales as Moderate; Grade 3 scales as severe or medically significant but not immediately life threatening; Grade 4 scales as life-threatening consequences; and Grade 5 scales as death related to AE.
Time Frame: From the start of the study drug up to Day 30 after the last dose of study drug (up to 8 months)
Population: as for outcome 11
Measure: Number; unit: percentage of participants
Arm/Group | Part 1, Sequence A: TAK-931 80 mg PIC + TAK-931 80 mg Tablet | Part 1, Sequence B: TAK-931 80 mg Tablet + TAK-931 80 mg PIC
Number analyzed (Participants) | 12 | 8
percentage of participants | 41.7 | 37.5

13. Secondary Outcome: Part 1: Percentage of Participants With Shift From Baseline Values to Post-baseline Values in Laboratory Parameters
Time Frame: From the start of the study drug up to Day 30 after the last dose of study drug (up to 8 months)
Population: as for outcome 11
Measure: Number; unit: percentage of participants
Arm/Group | Part 1, Sequence A: TAK-931 80 mg PIC + TAK-931 80 mg Tablet | Part 1, Sequence B: TAK-931 80 mg Tablet + TAK-931 80 mg PIC
Number analyzed (Participants) | 12 | 8
percentage of participants
  Eosinophils: Grade 0 to Grade 0 | 83.3 | 87.5
  Eosinophils: Grade 0 to Grade 1 | 8.3 | 0.0
  Eosinophils: Grade 1 to Grade 0 | 8.3 | 12.5
  Hemoglobin: Grade 0 to Grade 0 | 33.3 | 0.0
  Hemoglobin: Grade 0 to Grade 1 | 8.3 | 12.5
  Hemoglobin: Grade 1 to Grade 0 | 8.3 | 0.0
  Hemoglobin: Grade 1 to Grade 1 | 41.7 | 50.0
  Hemoglobin: Grade 1 to Grade 2 | 8.3 | 12.5
  Hemoglobin: Grade 1 to Grade 3 | 0.0 | 12.5
  Hemoglobin: Grade 2 to Grade 2 | 0.0 | 12.5
  Leukocytes: Grade 0 to Grade 0 | 41.7 | 75.0
  Leukocytes: Grade 0 to Grade 1 | 41.7 | 12.5
  Leukocytes: Grade 0 to Grade 2 | 16.7 | 0.0
  Leukocytes: Grade 0 to Grade 3 | 0.0 | 12.5
  Lymphocytes: Grade 0 to Grade 0 | 33.3 | 50.0
  Lymphocytes: Grade 0 to Grade 1 | 16.7 | 12.5
  Lymphocytes: Grade 0 to Grade 2 | 16.7 | 12.5
  Lymphocytes: Grade 0 to Grade 3 | 8.3 | 0.0
  Lymphocytes: Grade 1 to Grade 1 | 8.3 | 0.0
  Lymphocytes: Grade 1 to Grade 2 | 16.7 | 0.0
  Lymphocytes: Grade 2 to Grade 2 | 0.0 | 12.5
  Lymphocytes: Grade 3 to Grade 2 | 0.0 | 12.5
  Neutrophils: Grade 0 to Grade 0 | 83.3 | 75.0
  Neutrophils: Grade 0 to Grade 2 | 8.3 | 12.5
  Neutrophils: Grade 0 to Grade 3 | 8.3 | 0.0
  Neutrophils: Grade 0 to Grade 4 | 0.0 | 12.5
  Platelets: Grade 0 to Grade 0 | 100.0 | 62.5
  Platelets: Grade 0 to Grade 1 | 0.0 | 25.0
  Platelets: Grade 1 to Grade 1 | 0.0 | 12.5
  Alanine Aminotransferase: Grade 0 to Grade 0 | 91.7 | 62.5
  Alanine Aminotransferase: Grade 0 to Grade 1 | 0.0 | 25.0
  Alanine Aminotransferase: Grade 1 to Grade 0 | 8.3 | 0.0
  Alanine Aminotransferase: Grade 1 to Grade 1 | 0.0 | 12.5
  Alkaline Phosphatase: Grade 0 to Grade 0 | 33.3 | 0.0
  Alkaline Phosphatase: Grade 0 to Grade 1 | 16.7 | 37.5
  Alkaline Phosphatase: Grade 1 to Grade 0 | 33.3 | 25.0
  Alkaline Phosphatase: Grade 2 to Grade 0 | 8.3 | 37.5
  Alkaline Phosphatase: Grade 3 to Grade 0 | 8.3 | 0.0
  Aspartate Aminotransferase: Grade 0 to Grade 0 | 58.3 | 50.0
  Aspartate Aminotransferase: Grade 0 to Grade 1 | 25.0 | 0.0
  Aspartate Aminotransferase: Grade 1 to Grade 0 | 8.3 | 12.5
  Aspartate Aminotransferase: Grade 1 to Grade 1 | 8.3 | 25.0
  Aspartate Aminotransferase: Grade 2 to Grade 0 | 0.0 | 12.5
  Bilirubin: Grade 0 to Grade 0 | 83.3 | 87.5
  Bilirubin: Grade 0 to Grade 1 | 16.7 | 12.5
  Creatinine: Grade 0 to Grade 0 | 66.7 | 75.0
  Creatinine: Grade 0 to Grade 1 | 16.7 | 0.0
  Creatinine: Grade 0 to Grade 2 | 8.3 | 0.0
  Creatinine: Grade 1 to Grade 1 | 8.3 | 25.0
  Glucose: Grade 0 to Grade 0 | 100.0 | 100.0
  Magnesium: Grade 0 to Grade 0 | 50.0 | 50.0
  Magnesium: Grade 0 to Grade 1 | 8.3 | 25.0
  Magnesium: Grade 1 to Grade 1 | 41.7 | 25.0
  Potassium: Grade 0 to Grade 0 | 83.3 | 62.5
  Potassium: Grade 0 to Grade 1 | 8.3 | 12.5
  Potassium: Grade 0 to Grade 3 | 0.0 | 12.5
  Potassium: Grade 1 to Grade 1 | 8.3 | 12.5
  Sodium: Grade 0 to Grade 0 | 50.0 | 75.0
  Sodium: Grade 0 to Grade 1 | 41.7 | 25.0
  Sodium: Grade 1 to Grade 0 | 8.3 | 0.0

ADVERSE EVENTS:
Time Frame: TEAEs are adverse events (AE) that started after the first dose of study drug up to 30 days after the last dose of study drug (up to 8 months)
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment. As planned, safety data was collected and analyzed as per sequence and in accordance with the study design.
Arm/Group | Part 1, Sequence A: TAK-931 80 mg PIC + TAK-931 80 mg Tablet | Part 1, Sequence B: TAK-931 80 mg Tablet + TAK-931 80 mg PIC
All-Cause Mortality (participants affected / at risk) | 0/12 | 1/8
Serious Adverse Events (participants affected / at risk) | 2/12 | 2/8
Other Adverse Events (participants affected / at risk) | 9/12 | 6/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1, Sequence A: TAK-931 80 mg PIC + TAK-931 80 mg Tablet (N=12) | Part 1, Sequence B: TAK-931 80 mg Tablet + TAK-931 80 mg PIC (N=8)
Ileus (Gastrointestinal disorders) | 2 (3) | 0 (0)
Bundle branch block left (Cardiac disorders) | 0 (0) | 1 (1)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cholecystitis infective (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1, Sequence A: TAK-931 80 mg PIC + TAK-931 80 mg Tablet (N=12) | Part 1, Sequence B: TAK-931 80 mg Tablet + TAK-931 80 mg PIC (N=8)
Nausea (Gastrointestinal disorders) | 3 (3) | 4 (6)
Constipation (Gastrointestinal disorders) | 2 (2) | 4 (4)
Vomiting (Gastrointestinal disorders) | 2 (5) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (2) | 0 (0)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 6 (8) | 6 (10)
Oedema peripheral (General disorders) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 4 (7) | 2 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 1 (1) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 0 (0) | 1 (2)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 1 (1)
Otitis media (Infections and infestations) | 1 (2) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Rash pustular (Infections and infestations) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 1 (1)
Aphasia (Nervous system disorders) | 1 (1) | 0 (0)
Disturbance in attention (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Facial nerve disorder (Nervous system disorders) | 1 (1) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 1 (2)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Dry eye (Eye disorders) | 1 (1) | 1 (1)
Hepatic pain (Hepatobiliary disorders) | 1 (1) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Research Organization shall not publish any articles or papers nor make any presentations, nor assist any other person in publishing any articles or papers or in making any presentations relating or referring to the Study or any results, data or insights from or any data, information or materials obtained or generated in the performance of its obligations without the prior written consent of Takeda, which consent may be granted or withheld in Takeda's sole discretion.

DOCUMENTS (2):
  • Study Protocol (2018-06-21): https://cdn.clinicaltrials.gov/large-docs/11/NCT03708211/Prot_000.pdf
  • Statistical Analysis Plan (2020-03-05): https://cdn.clinicaltrials.gov/large-docs/11/NCT03708211/SAP_001.pdf